CLINICAL TRIAL: NCT00948467
Title: A Multicenter, Open-label, Dose-escalation, Phase I Study of TAK-733, an Oral MEK Inhibitor, in Adult Patients With Advanced Nonhematologic Malignancies
Brief Title: Study of TAK-733 in Adult Patients With Advanced Nonhematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C20001
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Advanced Non-hematologic Malignancies; Advanced Metastatic Melanoma
Keywords: Advanced nonhematologic malignancies; Advanced metastatic melanoma; BRAF gene
MeSH Terms: interventions — TAK 733

ARMS (1):
- TAK-733 (Experimental)
  Interventions: Drug: TAK-733

INTERVENTIONS:
Drug: TAK-733 — The Initial Escalation Stage will enroll approximately 30 patients with advanced nonhematologic malignancies. TAK-733 will be administered orally in 28-day treatment cycles consisting of intermittent dosing with 21 days of continuous treatment, followed by a rest period of 7 days.
  The Expansion Stage will enroll approximately 30 patients with advanced metastatic melanoma. The recommended phase 2 dose determined in the Initial Escalation Stage of TAK-733 will be administered orally in 28-day treatment cycles consisting of intermittent dosing with 21 days of continuous treatment, followed by a rest period of 7 days.

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, pharmacodynamics and maximum tolerated dose of TAK-733 in patients with advanced, nonhematologic tumors. The expansion stage of the study will evaluate evidence of antitumor activity of TAK-733 in patients with advanced metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* 18 years or older.
* Have one of the following diagnoses: a nonhematologic malignancy for which standard, curative, or life-prolonging treatment does not exist or is no longer effective; OR have stage 3 or stage 4 unresectable melanoma not priorly treated with either MEK or BRAF inhibitor therapy.
* Melanoma patients should have the V600E BRAF mutation status of their tumor documented, if available, and tumor tissue must be provided for confirmatory genotyping by a central laboratory.
* Have a radiographically or clinically evaluable tumor.
* Have suitable venous access for the conduct of blood sampling.
* Provide voluntary written consent, which can be withdrawn by the patient at any time.
* Female patients who: are post-menopausal for at least 1 year before screening; OR are surgically sterile; OR if they are of childbearing potential agree to practice two effective methods of birth control from the time of signing the informed consent form through 30 days after the last dose of the study drug, or agree to completely abstain from heterosexual intercourse.
* Male patients, even if surgically sterilized, must agree to practice effective barrier contraception during the entire study treatment period and through 30 days after the last dose of the study drug; OR agree to completely abstain from heterosexual intercourse.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Female patients who are lactating or have a positive serum pregnancy test during the Screening period.
* Antineoplastic therapy or radiotherapy within 21 days; or nitrosoureas of mitomycin C within 42 days
* Prior biologic or immunotherapy ≤ 4 weeks prior to enrollment.
* Grade 2 or greater unresolved toxicity (except alopecia) from previous anticancer therapy.
* Major surgery within 14 days of the first dose of the study drug.
* An active infection requiring systemic therapy; or other severe infection.
* Symptomatic brain metastases.
* Inability to meet specific laboratory test standards during the Screening period as specified in the study protocol.
* Human Immunodeficiency (HIV) positive.
* Hepatitis B surface antigen positive or active hepatitis C infection.
* Serious medical or psychiatric illness likely to interfere with the study.
* Uncontrolled cardiovascular condition.
* Abnormalities on 12-lead ECG performed within 28 days before the start of the study drug that are considered to be clinically significant or rate corrected QT interval > 470 milliseconds.
* Melanoma patients will be excluded if they have had a diagnosis with or treatment for another malignancy within 2 years of the first dose of the study drug, or have been previously diagnosed with another malignancy with any evidence of residual disease.
* Treatment with any investigational product within 28 days before the first dose of the study drug.
* A history of an ongoing or newly diagnosed eye abnormality, such as retinal or corneal pathologies.
* Abnormal left ventricular ejection fraction (LVEF).
* Receiving therapeutic anticoagulation
* Treatment with any of the following strong CYP3A inhibitors or inducers within 14 days before the first dose of study drug: ketoconazole, itraconazole, voriconazole, posaconazole, clarithromycin, telithromycin, nefazodone, rifampin, rifapentine, or rifabutin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-12; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety profile, dose-limiting toxicities, maximum tolerated dose and recommended phase 2 dose of TAK-733 | 12 months
Pharmacokinetic characterization of TAK-733 | 12 months

SECONDARY OUTCOMES:
Effect of food on the pharmacokinetics of TAK-733 | 12 months
Antitumor activity of TAK-733 in patients with advanced nonhematologic malignancies | 12 months
Antitumor activity of TAK-733 in melanoma patients | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Wayne State University Karmanos Cancer Institute, Detriot, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York